CLINICAL TRIAL: NCT07335237
Title: Objective: POGD is the Most Prevalent Complication Following Colon Cancer Surgery. The Integration of Acupuncture With ERAS Management Represents an Effective Approach for the Prevention and Treatment of POGD. Autonomic Nerve Function Serves as a Promising Target for Acupuncture Therapy; However, Its Precise Clinical Efficacy and Underlying Mechanisms Warrant Further Investigation. This Study Examines the Changes in Autonomic Nerve Function, Postoperative Gastrointestinal Recovery, and the Incidence of POGD in Patients Undergoing Colorectal Cancer Resection Under the ERAS Management Pathway, c
Brief Title: Clinical Study on the Prevention and Treatment of Postoperative Gastrointestinal Dysfunction by Acupuncture Under ERAS Management Based on Artificial Intelligence Monitoring
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Sun Wenhao, M.D., Jiangsu Province Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022NL-KS100
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Colectomy; Colectomy Left/Right/Total Under Laparotomy; Cancer; Chinese Medicine; Accupuncture; Heart Rate
Keywords: Colectal Cancer; Chinese Medicine; Accupuncture
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard ERAS Management (Active Comparator): Patients in this arm receive standard perioperative care following the established Enhanced Recovery After Surgery (ERAS) protocols, including early mobilization and early oral feeding, without acupuncture intervention.
  Interventions: Other: Accupuncture

INTERVENTIONS:
Other: Accupuncture — Specific Synergistic Acupoint Selection: The protocol uses a specialized combination of four acupoints-Zusanli (ST36), Neiguan (PC6), Tianshu (ST25), and Taichong (LR3). This specific "cluster" is designed not just for gut motility, but to specifically target the "Brain-Gut Axis" to reduce the systemic inflammatory response and postoperative pain simultaneously.
  High-Frequency Perioperative Timing: The intervention begins within 12 hours post-surgery, which is earlier than many traditional protocols. It is administered with a high-frequency density (every 12 hours for the first 72 hours), ensuring a consistent "dose" of neuro-stimulation during the most critical window of gastrointestinal paralysis.

SUMMARY:
Brief Summary: Acupuncture for Faster Recovery After Colorectal Surgery

1. What is this study about? Colorectal cancer is a common health condition that usually requires surgery. While surgery is effective, it often leads to a temporary "shutdown" of the digestive system, known as Postoperative Gastrointestinal Dysfunction (POGD). Patients may experience bloating, nausea, vomiting, and a delay in passing gas or having bowel movements. This study explores whether acupuncture can help the gut "wake up" faster and improve overall recovery.
2. Why is this research important? Currently, hospitals use a modern management system called ERAS (Enhanced Recovery After Surgery) to help patients recover. However, many patients still suffer from gut-related discomfort. We want to see if combining traditional Chinese medicine (acupuncture) with modern ERAS protocols provides a better, faster, and more comfortable recovery than ERAS alone.
3. What will happen during the study? Patients participating in this study at the affiliated hospital of Nanjing University of Chinese Medicine are randomly assigned to one of two groups:

   Standard Group: Receives standard ERAS care (early movement, early eating, and pain management).

   Acupuncture Group: Receives standard ERAS care plus professional acupuncture sessions.

   The Procedure: Fine, sterile needles are applied to specific points (such as Zusanli and Neiguan) for 30 minutes, twice a day for the first three days after surgery.

   Monitoring: To understand how the body responds, we use a non-invasive Artificial Intelligence (AI) monitor to track Heart Rate Variability (HRV). This helps us see how the nervous system is helping the gut recover in real-time.
4. What are the potential benefits? Based on our research findings involving 70 clinical cases, patients who received acupuncture experienced:

   Faster Recovery: The first passage of gas occurred approximately 23 hours earlier than those in the standard group.

   Shorter Hospital Stay: Patients were able to go home on average one day sooner.

   Less Pain: Acupuncture significantly reduced postoperative pain levels.

   Fewer Complications: A lower rate of severe digestive issues after surgery.
5. Is it safe? Acupuncture is a safe, drug-free, and minimally invasive therapy. It works by stimulating the vagus nerve and balancing the body's internal systems. Combined with the precision of AI monitoring, this approach ensures that the recovery process is both natural and scientifically tracked.
6. Conclusion The goal of this study is to provide a "green" and effective solution to help colorectal cancer patients suffer less after surgery and return to their normal lives as quickly as possible.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 80 years, male or female.
2. Diagnosed with colorectal malignancy by pathology or cytology.
3. Scheduled for elective radical resection of colorectal cancer (laparoscopic or open surgery).
4. ASA physical status classification: I-III.
5. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Patients with severe primary diseases of the heart, brain, kidney, hematopoietic, or endocrine systems.
2. History of major abdominal surgery or intestinal obstruction that significantly alters bowel anatomy.
3. Emergency surgery cases (e.g., acute obstruction, perforation, or peritonitis).
4. Contraindications to acupuncture (e.g., local skin infection, scars, or severe coagulation disorders).
5. Currently participating in other clinical trials.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Time to first postoperative flatus | From the end of surgery until the first passage of flatus, typically expected within 72 to 120 hours post-surgery.
  This measure records the duration (in hours) from the completion of the surgical procedure (end of skin closure) to the patient's first reported passage of flatus. It serves as a key clinical indicator of the recovery of intestinal motility and the resolution of postoperative ileus.

SECONDARY OUTCOMES:
Time to first postoperative defecation | From the end of the surgery until the 7th day after the operation (or until the patient is discharged from the hospital).
  Record the time elapsed from the end of the surgery (when the skin stitches were completed) until the patient passed their first stool after the operation, in hours. The occurrence of a bowel movement indicates the recovery of gastrointestinal motility.

CONTACTS AND LOCATIONS:
Locations (1):
- Affliated Hospital of Nanjing Universitty of Chinese Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided